CLINICAL TRIAL: NCT04153123
Title: Ophthalmic Artery Resistance Index After Peribulbar Block in the Presence of Epinephrine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Renato Santiago Gomez, Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CAAE 04433113.0.0000.5149
Record Dates: First submitted 2019-11-03; First posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Ophthalmic Artery; Peribulbar Block
Keywords: ocular flow; cataract surgery; peribulbar block; ocular Doppler
MeSH Terms: interventions — Epinephrine

STUDY DESIGN:
Intervention Model Description: Group 1: Peribulbar anesthesia with 2% lidocaine with epinephrine 1/200,000.
  Group 2: Peribulbar anesthesia with 2% lidocaine without epinephrine.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The preparation of the syringes was performed by one of the researchers not involved in the execution of the blockades. The same anesthesiologist performed all the blocks, while the same ophthalmologist did the ocular monitoring measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine with epinephrine (Experimental): Peribulbar anesthesia with lidocaine and epinephrine
  Interventions: Drug: Epinephrine
- Lidocaine without epinephrine (No Intervention): Peribulbar anesthesia with lidocaine

INTERVENTIONS:
Drug: Epinephrine
  Arms: Lidocaine with epinephrine

SUMMARY:
Evaluate ophthalmic artery flow by echo-Doppler before and after peribulbar block with lidocaine in presence or absence of epinephrine.

DETAILED DESCRIPTION:
There are controversies regarding the ophthalmic artery (OA) flow after peribulbar block with the addition of epinephrine. Therefore, we aimed to evaluate OA flow by echo-Doppler before and after peribulbar block with lidocaine in presence or absence of epinephrine.

Fifty-six patients that were eligible for cataract phacoemulsification surgery were selected. Patients were divided into two groups: group 1 - Peribulbar block with lidocaine and 1/200.000 epinephrine; group 2 - Peribulbar block with lidocaine in the absence of epinephrine. The resistance index (RI) of OA was evaluated using echo-Doppler before and 10 min after the peribulbar block.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I, II or III physical status classification
* Cataract surgery

Exclusion Criteria:

* glaucoma
* diabetic retinopathy
* previous eye surgery in the same eye
* ocular trauma
* allergic to any protocol medication
* uncooperative patients or cognitive difficulties
* axial eye diameter of less than 21.0 mm or greater than 25.5 mm.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2014-05-31 (Actual); Study Completion 2014-05-31 (Actual)

PRIMARY OUTCOMES:
Artery resistance index of ophthalmic artery | Change on resistance index 10 minutes after peribulbar anesthesia
  The resistance index (RI) of OA was evaluated using echo-Doppler before and 10 minutes after the peribulbar block.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Minas Gerais, Faculdade de Medicina, Departamento de Cirurgia., Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No
The data will be present at an official journal